CLINICAL TRIAL: NCT00877643
Title: Routine Versus Aggressive Upstream Rhythm Control for Prevention of Early Atrial Fibrillation in Heart Failure: RACE 3
Brief Title: Routine Versus Aggressive Upstream Rhythm Control for Prevention of Early Atrial Fibrillation in Heart Failure
Acronym: RACE 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.C. Van Gelder (Other)
Collaborators: The Interuniversity Cardiology Institute of the Netherlands (Other Government); Netherlands Heart Foundation (Other); Dutch Network for Cardiovascular Research (Unknown); Trial Coordination Center UMC Groningen (Unknown); Bayer (Industry); Boehringer Ingelheim (Industry); Medtronic (Industry); Biotronik SE & Co. KG (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, I.C. Van Gelder, Prof., University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHS B 2008 035; NHS B 2008 035
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upstream rhythm control (Experimental)
  Interventions: Other: Upstream therapy
- Conventional rhythm control (Active Comparator)
  Interventions: Other: Conventional rhythm control

INTERVENTIONS:
Other: Upstream therapy — Aldosterone receptor antagonists and statins, dietary restrictions, counseling, and cardiac rehabilitation.
  Arms: Upstream rhythm control
Other: Conventional rhythm control — Usual care for atrial fibrillation and heart failure according to the present guidelines
  Arms: Conventional rhythm control

SUMMARY:
The purpose of this study is to investigate whether in patients with early persistent atrial fibrillation and mild to moderate early heart failure an aggressive upstream rhythm control approach, including aldosterone receptor antagonists and statins, dietary restrictions, counseling and cardiac rehabilitation programs, increases persistence of sinus rhythm compared with conventional rhythm control after one year of follow-up.

A randomized long term extension of the RACE 3 will be performed with a total follow-up of 5 years to investigate the long term effects on persistence of sinus rhythm and cardiovascular morbidity and mortality of the two treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Early symptomatic persistent atrial fibrillation
* Mild to moderate early heart failure
* Optimal documentation and treatment of underlying heart disease
* No contra-indication for oral anticoagulation
* Eligible for cardiovascular rehabilitation
* Age >= 40 years

Exclusion Criteria:

* On waiting list for pulmonary vein isolation or expected to be placed on waiting list within one year
* Heart failure NYHA class IV
* LVEF < 25%
* Left atrial size > 50 mm (parasternal axis)
* Present aldosterone receptor antagonist use
* Previous use of class I or III antiarrhythmic drugs (except for sotalol, which should be discontinued at inclusion and replaced with betablocker)
* Cardiac resynchronization therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-05-04 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Success of rhythm control strategy consisting of 1) the patient is still in a rhythm control strategy according to the attending physician, and 2) that sinus rhythm is maintained after 1 year of follow-up. | 1 year after electrical cardioversion

SECONDARY OUTCOMES:
Exploratory randomized long term extension of the RACE 3 study performed to study the long term effects of the two treatment strategies. | 5 years after electrical cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alings, MD, PhD, Principal Investigator — Amphia Hospital Breda; Isabelle C Van Gelder, MD, PhD, Principal Investigator — University Medical Center Groningen; Harry J Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (20):
- Netherlands (15):
  - Ziekenhuisgroep Twente, Almelo
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Hospital Rijnstate, Arnhem
  - Ter Gooi Hospital, Blaricum
  - Amhia Hospital, Breda
  - Ommelander Hospital Group, Delfzijl
  - Deventer Hospital, Deventer
  - Oosterscheldeziekenhuis, Goes
  - Martini Hospital, Groningen
  - University Medical Center Groningen, Groningen
  - Kennemer Gasthuis, Haarlem
  - Medical University Center Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - Viecuri Hospital, Venlo
  - Ommelander Hospital Group, Winschoten
- United Kingdom (5):
  - City Hospital (Sandwell and West Birmingham Hospitals NHS Trust), Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Poole Hospital NHS Foundation Trust, Poole
  - Good Hope Hospital (Heart of England NHS Foundation Trust), Sutton Coldfield

REFERENCES:
- [Derived] Nguyen BO, Crijns HJGM, Tijssen JGP, Geelhoed B, Hobbelt AH, Hemels MEW, Mol WJM, Weijs B, Alings M, Smit MD, Tieleman RG, Tukkie R, Van Veldhuisen DJ, Van Gelder IC, Rienstra M; RACE 3 Investigators. Long-term outcome of targeted therapy of underlying conditions in patients with early persistent atrial fibrillation and heart failure: data of the RACE 3 trial. Europace. 2022 Jul 15;24(6):910-920. doi: 10.1093/europace/euab270. PMID 34791160
- [Derived] Nguyen BO, Rienstra M, Hobbelt AH, Tijssen JGP, Smit MD, Tieleman RG, Geelhoed B, Van Veldhuisen DJ, Crijns HJGM, Van Gelder IC; RACE 3 Investigators. Optimal treatment of underlying conditions improves rhythm control outcome in atrial fibrillation - Data from RACE 3. Am Heart J. 2020 Aug;226:235-239. doi: 10.1016/j.ahj.2019.12.005. Epub 2020 Feb 14. No abstract available. PMID 32067695
- [Derived] De With RR, Rienstra M, Smit MD, Weijs B, Zwartkruis VW, Hobbelt AH, Alings M, Tijssen JGP, Brugemann J, Geelhoed B, Hillege HL, Tukkie R, Hemels ME, Tieleman RG, Ranchor AV, Van Veldhuisen DJ, Crijns HJGM, Van Gelder IC. Targeted therapy of underlying conditions improves quality of life in patients with persistent atrial fibrillation: results of the RACE 3 study. Europace. 2019 Apr 1;21(4):563-571. doi: 10.1093/europace/euy311. PMID 30629160
- [Derived] Rienstra M, Hobbelt AH, Alings M, Tijssen JGP, Smit MD, Brugemann J, Geelhoed B, Tieleman RG, Hillege HL, Tukkie R, Van Veldhuisen DJ, Crijns HJGM, Van Gelder IC; RACE 3 Investigators. Targeted therapy of underlying conditions improves sinus rhythm maintenance in patients with persistent atrial fibrillation: results of the RACE 3 trial. Eur Heart J. 2018 Aug 21;39(32):2987-2996. doi: 10.1093/eurheartj/ehx739. PMID 29401239